CLINICAL TRIAL: NCT02123641
Title: Physical Activity as Intervention Against Age-related Loss of Muscle Mass and Function
Acronym: LISA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Michael Kjaer, Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: H-3-2014-017
Record Dates: First submitted 2014-04-24; First posted 2014-04-25 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Muscle Weakness; Muscle Loss; Sarcopenia; Physical Activity
MeSH Terms: conditions — Muscle Weakness; Muscular Atrophy; Sarcopenia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Heavy resistance training (Active Comparator): Heavy resistance training of the lower and upper extremities three times weekly for 52 weeks.
  Interventions: Other: Heavy resistance training
- Moderate intensity training (Experimental): Home-based moderate intensity training of the lower and upper extremities three times weekly for 52 weeks.
  Interventions: Other: Moderate intensity training
- Control (Experimental): No training
  Interventions: Other: Control

INTERVENTIONS:
Other: Heavy resistance training — Supervised heavy resistance training three times weekly for 52 weeks.
  Arms: Heavy resistance training
Other: Moderate intensity training — Moderate intensity training supervised once weekly and home based unsupervised two times weekly for 52 weeks.
  Arms: Moderate intensity training
Other: Control — No training
  Arms: Control

SUMMARY:
A minimum of 450 healthy individuals (62-70 years old) will be recruited.

Each individual will be randomized into one of three groups stratified according to gender (M/F), BMI (≤28/>28), and 30 sec chair stand (≤11/>11). The three groups are Heavy resistance training (n=150), moderate intensity training (n=150), and control (n=150, no training).

Assessments will be performed at baseline, after 12 months of intervention. Furthermore, follow up will be performed after 2,4,7, and 10 years.

The primary outcome is change in leg extensor power after the intervention and during follow up.

The primary hypothesis is that by applying the intention-to-treat analysis, the moderate intensity training group will increase leg extensor power just as much as the heavy resistance training group. The two training groups will increase muscle power more than the control group.

DETAILED DESCRIPTION:
Retirement has been recognized as a critical turning point in determining physical activity behaviours in old age. The literature gives a varying picture regarding change in physical activity level with work retirement but often a reduction in total physical activity has been reported. Retirement typically takes place at a time where the skeletal muscle mass, -strength and -power declines by 1-3% per year.

Interventions to promote physical activity in adults aged 55 to 70 years have been shown to be effective at 12 months but it is very unclear if the effect is maintained thereafter. Both exercise at home or at a center improves health and physical function - but home based programs appear to be superior to center based programs in terms of adherence to exercise especially in the long-term.

In older adults, strength training at 60% of 1RM has been shown to be sufficient for large effect on muscle function and muscle protein synthesis, and potentially lower loads (45-60% 1RM) have effect when adding more repetitions.

The overall objective of the study is to assess the long-term effects of 12 month of supervised high-intensity center based resistance training or "guided" moderate-intensity home-based resistance training relative to a non-exercising control group upon muscle power, -strength and -mass, physical function, physical activity level and health in older people around the time of retirement.

The hypotheses are:

1. Supervised high-intensity center based resistance training over one year results in the best improvement in muscle power and bodily function
2. "Guided" moderate-intensity home-based resistance training will result in a more active lifestyle and thus in sustained elevated activity level after the 1-year intervention period. Thus in the long run (several years) "guided" moderate-intensity home-based resistance training has superior effects compared to supervised high-intensity center based resistance training upon functional ability, health and potentially also cognitive function.

450 participants recruited through advertisements in local newspapers will be included in this three-armed, single-blinded randomized trial. After baseline assessment they will be randomized to one year of 1) supervised, high-intensity progressive, resistance training conducted in machines three times weekly in a local fitness center 2) "guided" moderate-intensity home-based resistance training conducted with elastic bands and body weight three times weekly. "Guided" means that the participants are offered supervised resistance training once weekly in addition to home based resistance training 2 times weekly or 3) various social and cultural activities that do not require physical activity.

All participants complete a wide range of tests before and after the 12 months intervention period and the primary time point for outcome assessment will be at 12 month. The same "test battery" is conducted in the subsequent years (2, 4, 7, and 10 years later) as a follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Independently living men and women
* Between 62 and 70 years

Exclusion Criteria:

* Subjects dependent on help/nursing etc.
* Severe chronic obstructive pulmonary disease, cardiac arrhythmias or known decreased left ventricular ejection fraction, non-treated hyper/hypothyroidism, dementia, active cancer.
* Surgical diseases: Bone, muscle, tendon or joint injuries compromising participation in exercise regimens.
* Implanted magnetic devices incompatible with MRi-scanning.
* >1 hour of exercise weekly, except light activities such as stretching/gymnastics and bike-riding/walking as transportation.

Ages: 62 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2014-04; Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change in leg extensor power | Baseline, 1, 2, 4, 7, and 10 years follow up
  Unilateral leg extension power measured in the Leg Extensor Power Rig device (Nottingham). The primary time interval for assessment of the primary outcome measure is from baseline to 12 months intervention. The statistical evaluation of the primary outcome measure is done by applying a two way ANOVA test comparing the three groups before/after the intervention and during follow up (1,2,4,7, and 10 years).

SECONDARY OUTCOMES:
Change in quadriceps cross sectional area | Baseline, 1, 2, 4, 7, and 10 years
  MRI scanning of thigh muscle composition
Change in maximal isometric quadriceps strength | Baseline, 1, 2, 4, 7, and 10 years
  Unilateral maximal isometric quadriceps strength measured in the Good Strength device.
Change in 30 s chair stand performance | Baseline, 1, 2, 4, 7, and 10 years
  Number of stand-ups from a chair in 30 seconds
Change in 400 m gait speed | Baseline, 1, 2, 4, 7, and 10 years
  The time used for walking 400 m (20 m course)
Change in whole body composition and bone mineral density as well as lumbar spine and femoral neck bone mineral density | Baseline, 1, 2, 4, 7, and 10 years
  Body composition (fat mass, lean mass and bone mass) evaluated by whole-body and regional (lumbar spine and femoral neck) dual energy x-ray absorptiometry (DXA)-scanning.
Change in grip strength | Baseline, 1, 2, 4, 7, and 10 years
  Isometric hand grip strength (Saehan dynamometer)
Change in perceived age | Baseline, 1, 2, 4, 7, and 10 years
  Determination of perceived age from facial and whole-body photographs
Change in blood parameters and anthropometry | Baseline, 1, 2, 4, 7, and 10 years
  Measuring 1) blood levels of inflammatory markers (CRP, TNFa, and IL-6) and HbA1c, plasma lipids. 2) Weight, abdominal circumference, blood pressure.
Change in physical activity level | Baseline, 1, 2, 4, 7, and 10 years
  Wearing a pedometer device (ActivPal) for 5 continuous days. Questionnaire: PASE (Physical Activity Scale for the Elderly).
Change in Exercise self-efficacy | Baseline, 1, 2, 4, 7, and 10 years
  Questionnaire: Exercise Self-efficacy Scale.
Change in Health Related Quality of Life | Baseline, 1, 2, 4, 7, and 10 years
  Questionnaire: SF36.
Changes in brain structure and function | Baseline, 1, 2, 4, 7, and 10 years
  MRI scanning of the regional brain structure and function
Change in cognitive ability | Baseline, 1, 2, 4, 7, and 10 years
  Questionnaire: IST 2000-R
Change in personality | Baseline, 1, 2, 4, 7, and 10 years
  Questionnaire: NEO-FFI
Change in mental symptoms | Baseline, 1, 2, 4, 7, and 10 years
  Questionnaire: SCL-90
Adherence to training interventions | 2, 4, 7, 10 years
  Questionnaire developped specifically for the LISA study by the authores

CONTACTS AND LOCATIONS:
Overall Officials: Kasper Dideriksen, PhD stud, Principal Investigator — Bispebjerg Hospital; Anne Gylling, PhD stud, Principal Investigator — Bispebjerg Hospital; Christian Eriksen, PhD stud, Principal Investigator — Bispebjerg Hospital; Michael Kjaer, MD, Proff, Principal Investigator — Bispebjerg Hospital; Andreas Ziegler, PhD stud, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bloch-Ibenfeldt M, Demnitz N, Gates AT, Garde E, Siebner HR, Kjaer M, Boraxbekk CJ. No long-term benefits from resistance training on brain grey matter volumes in active older adults at retirement age. BMC Geriatr. 2025 Feb 21;25(1):120. doi: 10.1186/s12877-025-05778-z. PMID 39984875
- [Derived] Bloch-Ibenfeldt M, Gates AT, Jorgensen NR, Linneberg A, Aadahl M, Kjaer M, Boraxbekk CJ. Heavy resistance training provides short-term benefits on bone formation in well-functioning older adults. Bone. 2025 Apr;193:117393. doi: 10.1016/j.bone.2025.117393. Epub 2025 Jan 18. PMID 39832659
- [Derived] Bloch-Ibenfeldt M, Theil Gates A, Karlog K, Demnitz N, Kjaer M, Boraxbekk CJ. Heavy resistance training at retirement age induces 4-year lasting beneficial effects in muscle strength: a long-term follow-up of an RCT. BMJ Open Sport Exerc Med. 2024 Jun 18;10(2):e001899. doi: 10.1136/bmjsem-2024-001899. eCollection 2024. PMID 38911477
- [Derived] Gylling AT, Eriksen CS, Garde E, Wimmelmann CL, Reislev NL, Bieler T, Ziegler AK, Andersen KW, Bauer C, Dideriksen K, Baekgaard M, Mertz KH, Bayer ML, Bloch-Ibenfeldt M, Boraxbekk CJ, Siebner HR, Mortensen EL, Kjaer M. The influence of prolonged strength training upon muscle and fat in healthy and chronically diseased older adults. Exp Gerontol. 2020 Jul 15;136:110939. doi: 10.1016/j.exger.2020.110939. Epub 2020 Apr 8. PMID 32277977
- [Derived] Modig K, Talback M, Ziegler L, Ahlbom A. Temporal trends in incidence, recurrence and prevalence of stroke in an era of ageing populations, a longitudinal study of the total Swedish population. BMC Geriatr. 2019 Feb 4;19(1):31. doi: 10.1186/s12877-019-1050-1. PMID 30717697
- [Derived] Eriksen CS, Svensson RB, Gylling AT, Couppe C, Magnusson SP, Kjaer M. Load magnitude affects patellar tendon mechanical properties but not collagen or collagen cross-linking after long-term strength training in older adults. BMC Geriatr. 2019 Jan 31;19(1):30. doi: 10.1186/s12877-019-1043-0. PMID 30704412
- [Derived] Eriksen CS, Garde E, Reislev NL, Wimmelmann CL, Bieler T, Ziegler AK, Gylling AT, Dideriksen KJ, Siebner HR, Mortensen EL, Kjaer M. Physical activity as intervention for age-related loss of muscle mass and function: protocol for a randomised controlled trial (the LISA study). BMJ Open. 2016 Dec 2;6(12):e012951. doi: 10.1136/bmjopen-2016-012951. PMID 27913559